CLINICAL TRIAL: NCT06406322
Title: Effects of Aerobic Exercise Training in Addition to Pelvic Floor Muscle Training in Gynecological Cancer Survivors With Pelvic Floor Dysfunction
Brief Title: Pelvic Floor Dysfunction and Aerobic Training in Gynecological Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Fatma Busra Benguboz, Lecturer, Atılım University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-BENGUBOZ-002
Record Dates: First submitted 2024-04-22; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Gynecologic Cancer; Pelvic Floor Disorders; Aerobic Exercise
Keywords: Pelvic Floor Dysfunction; Gynecologic Cancer; Physiotherapy
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Muscle Training (PFMT) Group (Active Comparator): Training will be planned for patients, including strengthening and endurance exercises,
  Interventions: Other: PFMT
- PFMT + Aerobic Exercise Group (Experimental): Both groups will be given PFMT, and the Grup B group will be given aerobic exercise training in addition to PFMT.
  Interventions: Other: PFMT; Other: Aerobic Exercise

INTERVENTIONS:
Other: PFMT — Pelvic floor muscle training will be given to patients with strengthening and endurance exercises for 8 weeks. PFMT will be applied at a patient-specific progression for 8 weeks.Exercises will be given in different positions (supine, sitting, etc.).
Other: Aerobic Exercise — Aerobic exercise will be applied as a progressive program in the form of a walking program, at least 4 days a week for 8 weeks. There will be 5-minute warm-up and cool-down periods (walking at a light pace) before and after exercise.
  Arms: PFMT + Aerobic Exercise Group

SUMMARY:
The incidence of gynecological cancer and the related death rates in the world are increasing every year. Unfortunately, pelvic floor disorders (PFDs) such as pelvic pain, dyspareunia, vaginal stenosis, and urinary incontinence can result from specific cancer treatments.

Our aim in our study is to examine the effects of aerobic exercise training in addition to pelvic floor muscle training on pelvic floor dysfunction symptoms, pelvic floor muscle strength and endurance, quality of life, functional capacity and fatigue in women surviving gynecological cancer with pelvic floor dysfunction.

Patients diagnosed with gynecological cancer and undergoing treatment will be invited to our research. Patients who meet the inclusion criteria and agree to participate will be divided into two groups as Pelvic Floor Muscle Training (PFMT) and PFMT+Aerobic Exercise by block randomization method.

For evaluation,We will use the Pelvic Floor Distress Inventory (PTDE-20), Pelvic Floor Impact Scale with digital palpation, EORTC QLQ-C30, 6 Minute Walk Test and Piper Fatigue Scale.

DETAILED DESCRIPTION:
Pelvic floor muscle training (PFMT) is recommended as a first-line conservative treatment in women with PFD. The purpose of these exercises is to maintain and improve pelvic floor muscle strength, endurance, flexibility, and coordination. In a study examining the effects of a home-based rehabilitation program on UI in endometrial cancer survivors, 12 weeks of PFMT, bladder, and life changes education were provided. As a result of the study, it was reported that the home program could be effective in reducing UI symptoms.

Aerobic exercise training is a method that can ameliorate the loss of skeletal muscle mass and function. In studies evaluating the relationship between physical activity and UI, there are studies showing that walking is positively associated with the reduction of UI symptoms. However, when the literature was examined, no study was found evaluating the effect of aerobic exercise training on PFD in individuals with gynecological cancer.

There are studies in the literature examining the effect of PFMT on different types of gynecological cancer. Studies have shown that different exercise programs are effective in reducing symptoms of pelvic floor dysfunctions seen after treatment in gynecological cancer patients and increasing pelvic floor muscle strength, thus increasing the quality of life. When the studies were examined, no study was found examining the effects of aerobic exercise training in addition to pelvic floor muscle training on PFD symptoms, pelvic floor muscle functions, quality of life, functional capacity, and fatigue in women surviving gynecological cancer.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who have at least one symptom of PFD (UI, anal incontinence, pelvic organ prolapse) due to gynecological cancer treatment,
* At least 12 months have passed since completing surgery, chemotherapy, or radiotherapy treatments,
* Being over 18 years old,
* Karnofsky performance scale being greater than 90,
* Being literate.

Exclusion Criteria:

* Having symptoms of pelvic floor dysfunction before cancer diagnosis,
* Diagnosed with metastatic cancer,
* Having a pelvic infection,
* Having any orthopedic, neurological, or cardiopulmonary disease that would prevent them from exercising,
* Having morbid obesity,
* Those who have communication and cooperation problems.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Symptoms | change from baseline at 8 weeks
  The Pelvic Floor Distress Inventory (PFDI-20) will be used to measure the severity of patients' pelvic floor symptoms.The PFDI-20 scale consists of 20 questions in total and three subscales: Urinary Distress Inventory (UDI-6), Pelvic Organ Prolapse Distress Inventory (POPDI-6), and Colorectal-Anal Distress Inventory (CRADI-8) .A total of 0-300 points can be obtained in the three sections. As the score approaches 300, the degree of complaint increases.

SECONDARY OUTCOMES:
Pelvic floor muscle strength | change from baseline at 8 weeks
  Pelvic floor muscle strength will be assessed during digital palpation with the Modified Oxford Scale (MOS) . Scoring according to squeezing intensity is done and noted as follows: 0 = No contraction, 1 = Very weak, 2 = Weak, 3 = Moderate, 4 = Good, and 5 = Strong. During the evaluation by digital palpation, the duration of contraction for muscle endurance will also be recorded.
Quality of life due to pelvic floor dysfunctions | change from baseline at 8 weeks
  The Pelvic Floor Impact Scale-7 will be used to evaluate patients' quality of life due to pelvic floor dysfunctions. The scale is a functional status measure that evaluates the impact of a person's bowel, bladder, and/or pelvic symptoms on different daily living activities, social relationships, or emotions. A scale score between 0 and 100 is obtained for each subscale. A high score indicates poor quality of life.
Cancer-related quality of life | change from baseline at 8 weeks
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) will be used to evaluate patients' cancer-related quality of life. The scale consists of three subheadings: general well-being, functional area, and symptom control. While high scores for all sections except the symptom score indicate a high quality of life, high scores for the symptom score indicate low quality of life.
Functional capacity | change from baseline at 8 weeks
  To evaluate functional capacity, patients will undergo a 6-minute walk test (6MWT) in accordance with the American Thoracic Society criteria. Individuals will be asked to walk at their maximum speed along a 30-meter corridor. The distance walked by the patient until the time is up or the point they wish to finish the test will be recorded.
Fatigue | change from baseline at 8 weeks
  Functional Assessment in the Treatment of Chronic Diseases - Fatigue Scale will be used to evaluate patients' fatigue.The scores that can be obtained from the scale vary between 0-52. A high total score on the scale indicates that the severity of fatigue is low.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda TOPRAK CELENAY, Assoc. Prof., Study Chair — Ankara Yildirim Beyazıt University